CLINICAL TRIAL: NCT04964830
Title: Sleep, Upper Airway and Dental Occlusion in Children With Large Overjet Before and After Treatment With a Mandibular Advancement Device (MAD)
Brief Title: Sleep, Upper Airway and Dental Occlusion in Children With Large Overjet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Postgraduate Programme in Orthodontics, Copenhagen (Unknown); Sygekassernes Helsefond (Other); The Danish Dental Association (Unknown); Københavns Kommune (Other); Hørsholm Kommune (Unknown); Rødovre Kommune (Unknown); Hvidovre Kommune (Unknown); Høje-Taastrup Kommune (Unknown)
Responsible Party: Principal Investigator, Camilla Hansen, PhD student, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-17011521
Record Dates: First submitted 2021-06-01; First posted 2021-07-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Overjet, Dental
Keywords: sleep; upper airway; dental occlusion; jaw function; overjet; children; adolescents
MeSH Terms: conditions — Overbite; Bites and Stings | interventions — Orthodontics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with large overjet (Active Comparator): Overjet ≥6 mm, planned orthodontic treatment with functional appliance
  Interventions: Device: Orthodontic treatment with functional appliance (MAD)
- Control group (No Intervention): Neutral occlusion, no indication for orthodontic treatment, no prior orthodontic treatment

INTERVENTIONS:
Device: Orthodontic treatment with functional appliance (MAD) — Expansion plate and z-activator (MAD)
  Arms: Children with large overjet

SUMMARY:
This project examines sleep (e.g. prevalence of obstructive sleep apnea(OSA)), dimension of upper airway, jaw function, well-being and quality of life in children with large overjet compared to a control group. In addition, the effect of treatment with a mandibular advancement device (MAD) on sleep, upper airway and jaw function are examined, and how these factors affect the children's well-being and quality of life.

DETAILED DESCRIPTION:
Sleep is very important for children's growth, development and learning. The anatomy and size of the airway and position of the jaw can affect children's sleep. Children with large overjet due to a posterior position of the mandible have smaller airways compared to children with neutral occlusion. Reduced dimensions of the upper airways may increase the risk of impaired sleep quality and the sleep related breathing disorder obstructive sleep apnoea (OSA), which causes symptoms e.g. failure to thrive, irritability, behavioural disorders, fatigue, which affects the children's growth, development, and learning negatively.

Children with large overjet due to mandibular retrognathia in Denmark are offered orthodontic treatment in municipal dental care and are in most cases treated with a mandibular advancement device (MAD) keeping the mandible in a forward position relative to the maxilla. MADs are also used to treat adults with mild-moderate obstructive sleep apnoea while they sleep. This can reduce the number of apnoea periods by up to 75% as well as preventing daytime sleepiness.

No previous study have examined sleep, upper airway, jaw function, well-being and quality of life in children with large overjet before, during and after MAD treatment compared to a control group with normal occlusion.

ELIGIBILITY:
Inclusion Criteria:

Overjet group:

* Horizontal maxillary overjet ≥ 6 mm and need of orthodontic treatment according to the Danish procedure for screening the child population for malocclusion involving health risk.
* Informed consent from parent(s)/guardian(s)

Control group:

* Neutral occlusion
* No history of orthodontic treatment
* Informed consent from parent(s)/guardian(s)

Exclusion Criteria:

* Known general and/or craniofacial syndromes/diseases
* Known sleep disorders, included bruxism during sleep
* Chronic respiratory diseases and asthma6/12
* Adenoid vegetations, hypertrophic tonsils and significantly reduces airflow through the nose (mouth breather), which need primary treatment.
* Dysfunction of masticatory muscles and temporomandibular joint, which need primary treatment.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence and grade of obstructive sleep apnea | Baseline
  Overnight polygraphy performed at home. Apnea: Reduction of ≥ 90 % of the oronasal airflow compared to baseline lasting for more than two breaths' duration.
  Hypopnea: Reduction of oronasal airflow of ≥ 30 % compared to baseline; desaturation of blood oxygen of ≥ 3% lasting for more than two breaths' duration, or association of desaturation with an arousal.
  Apnea-hypopnea pr hour during sleep (AHI-index) Normal: AHI <1; mild: AHI>1; moderate: AHI>5; severe: AHI>10
Presence and grade of obstructive sleep apnea | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Apnea: Reduction of ≥ 90 % of the oronasal airflow compared to baseline lasting for more than two breaths' duration.
  Hypopnea: Reduction of oronasal airflow of ≥ 30 % compared to baseline; desaturation of blood oxygen of ≥ 3% lasting for more than two breaths' duration, or association of desaturation with an arousal.
  Apnea-hypopnea pr hour during sleep (AHI-index) Normal: AHI <1; mild: AHI>1; moderate: AHI>5; severe: AHI>10
Presence and grade of obstructive sleep apnea | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Apnea: Reduction of ≥ 90 % of the oronasal airflow compared to baseline lasting for more than two breaths' duration.
  Hypopnea: Reduction of oronasal airflow of ≥ 30 % compared to baseline; desaturation of blood oxygen of ≥ 3% lasting for more than two breaths' duration, or association of desaturation with an arousal.
  Apnea-hypopnea pr hour during sleep (AHI-index) Normal: AHI <1; mild: AHI>1; moderate: AHI>5; severe: AHI>10
Oxygen desaturation index (ODI) | Baseline
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %. ODI is the number of desaturation events (a 4% decrease in SpO2%) per hour of total sleep ODI<1 is considered normal.
Oxygen desaturation index (ODI) | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %. ODI is the number of desaturation events (a 4% decrease in SpO2%) per hour of total sleep ODI<1 is considered normal.
Oxygen desaturation index (ODI) | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %. ODI is the number of desaturation events (a 4% decrease in SpO2%) per hour of total sleep ODI<1 is considered normal.
Snore Index | Baseline
  Overnight polygraphy performed at home. Snore Index %= time spent snoring / total time spent in bed.
Snore Index | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Snore Index %= time spent snoring / total time spent in bed.
Snore Index | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Snore Index %= time spent snoring / total time spent in bed.
Lowest SpO2% | Baseline
  Overnight polygraphy performed at home. The lowest value of oxygen saturation (SpO2%) measured in %; the optimal values are 94-100% Normal: SpO2% =92-100%; mild: SpO2% =89-91%; moderate: SpO2% =76-85%; severe: SpO2% =≤75%
Lowest SpO2% | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. The lowest value of oxygen saturation (SpO2%) measured in %; the optimal values are 94-100% Normal: SpO2% =92-100%; mild: SpO2% =89-91%; moderate: SpO2% =76-85%; severe: SpO2% =≤75%
Lowest SpO2% | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. The lowest value of oxygen saturation (SpO2%) measured in %; the optimal values are 94-100% Normal: SpO2% =92-100%; mild: SpO2% =89-91%; moderate: SpO2% =76-85%; severe: SpO2% =≤75%
Average SpO2% | Baseline
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %; the optimal values are 94-100% Normal: SpO2% =92-100%; mild: SpO2% =89-91%; moderate: SpO2% =76-85%; severe: SpO2% =≤75%
Average SpO2% | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %; the optimal values are 94-100% Normal: SpO2% =92-100%; mild: SpO2% =89-91%; moderate: SpO2% =76-85%; severe: SpO2% =≤75%
Average SpO2% | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %; the optimal values are 94-100% Normal: SpO2% =92-100%; mild: SpO2% =89-91%; moderate: SpO2% =76-85%; severe: SpO2% =≤75%
SpO2 under 90 % | Baseline
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %; the optimal values are 94-100%
SpO2 under 90 % | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %; the optimal values are 94-100%
SpO2 under 90 % | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Oxygen saturation (SpO2%) measured in %; the optimal values are 94-100%
Pulse Average | Baseline
  Overnight polygraphy performed at home. Average of the pulse during the total sleep Continuous scale
Pulse Average | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Average of the pulse during the total sleep Continuous scale
Pulse Average | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Average of the pulse during the total sleep Continuous scale
Oximeter quality % | Baseline
  Overnight polygraphy performed at home. Oximeter signal quality in % from 0-100.
  ≥75 % is considered good
Oximeter quality % | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Oximeter signal quality in % from 0-100.
  ≥75 % is considered good
Oximeter quality % | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Oximeter signal quality in % from 0-100.
  ≥75 % is considered good
Flow quality % | Baseline
  Overnight polygraphy performed at home. Nasal cannula flow signal quality in % from 0-100.
  ≥75 % is considered good
Flow quality % | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Nasal cannula flow signal quality in % from 0-100.
  ≥75 % is considered good
Flow quality % | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Nasal cannula flow signal quality in % from 0-100.
  ≥75 % is considered good
Respiratory inductance plethysmography (RIP) quality % | Baseline
  Overnight polygraphy performed at home. Thoracic and abdominal signal quality in % from 0-100.
  ≥75 % is considered good
Respiratory inductance plethysmography (RIP) quality % | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Thoracic and abdominal signal quality in % from 0-100.
  ≥75 % is considered good
Respiratory inductance plethysmography (RIP) quality % | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Thoracic and abdominal signal quality in % from 0-100.
  ≥75 % is considered good
Estimated sleep efficiency % | Baseline
  Overnight polygraphy performed at home. The percentage of time the child/adolescent sleep, in relation to the amount of time he/she spends in bed.
  Estimated sleep efficiency % = Total Sleep Time / Total Time in bed.
  ≥80 % is considered good/normal
Estimated sleep efficiency % | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. The percentage of time the child/adolescent sleep, in relation to the amount of time he/she spends in bed.
  Estimated sleep efficiency % = Total Sleep Time / Total Time in bed.
  ≥80 % is considered good/normal
Estimated sleep efficiency % | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. The percentage of time the child/adolescent sleep, in relation to the amount of time he/she spends in bed.
  Estimated sleep efficiency % = Total Sleep Time / Total Time in bed.
  ≥80 % is considered good/normal
Respiration rate | Baseline
  Overnight polygraphy performed at home. Number of breaths per minute Normal values according to age: 18-30 (6-12 years) and 12-20 (<12 years)
Respiration rate | 4-8 months from baseline (after expansion plate)
  Overnight polygraphy performed at home. Number of breaths per minute Normal values according to age: 18-30 (6-12 years) and 12-20 (<12 years)
Respiration rate | 14-18 months from baseline (after z-activator (MAD))
  Overnight polygraphy performed at home. Number of breaths per minute Normal values according to age: 18-30 (6-12 years) and 12-20 (<12 years)
Epworth Sleepiness Scale for Children and Adolescents (ESS(CHAD)) | Baseline
  ESS(CHAD) questionnaire: "Over the last month, how likely have you been to fall asleep while doing the listed activities?" Scale: 0 = would never fall asleep; 1 = slight chance of falling asleep; 2 = moderate chance of falling asleep; 3 = high chance of falling asleep.
  Interpretation of score: 0-5 Lower Normal Daytime Sleepiness; 6-10 Higher Normal Daytime Sleepiness; 11-12 Mild Excessive Daytime Sleepiness; 13-15 Moderate Excessive Daytime Sleepiness; 16-24 Severe Excessive Daytime Sleepiness.
Epworth Sleepiness Scale for Children and Adolescents (ESS(CHAD)) | 4-8 months from baseline (after expansion plate)
  ESS(CHAD) questionnaire: "Over the last month, how likely have you been to fall asleep while doing the listed activities?" Scale: 0 = would never fall asleep; 1 = slight chance of falling asleep; 2 = moderate chance of falling asleep; 3 = high chance of falling asleep.
  Interpretation of score: 0-5 Lower Normal Daytime Sleepiness; 6-10 Higher Normal Daytime Sleepiness; 11-12 Mild Excessive Daytime Sleepiness; 13-15 Moderate Excessive Daytime Sleepiness; 16-24 Severe Excessive Daytime Sleepiness.
Epworth Sleepiness Scale for Children and Adolescents (ESS(CHAD)) | 14-18 months from baseline (after z-activator (MAD))
  ESS(CHAD) questionnaire: "Over the last month, how likely have you been to fall asleep while doing the listed activities?" Scale: 0 = would never fall asleep; 1 = slight chance of falling asleep; 2 = moderate chance of falling asleep; 3 = high chance of falling asleep.
  Interpretation of score: 0-5 Lower Normal Daytime Sleepiness; 6-10 Higher Normal Daytime Sleepiness; 11-12 Mild Excessive Daytime Sleepiness; 13-15 Moderate Excessive Daytime Sleepiness; 16-24 Severe Excessive Daytime Sleepiness.
Berlin questionnaire | Baseline
  The questionnaire consists of 2 categories related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories 1 and 2.
  Category 1: 5 questions. Positive score if ≥2 points Category 2: 3 questions. Positive score if ≥2 points High Risk: if there are 2 or more categories where the score is positive. Low Risk: if there is only 1 or no categories where the score is positive.
Berlin questionnaire | 4-8 months from baseline (after expansion plate)
  The questionnaire consists of 2 categories related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories 1 and 2.
  Category 1: 5 questions. Positive score if ≥2 points Category 2: 3 questions. Positive score if ≥2 points High Risk: if there are 2 or more categories where the score is positive. Low Risk: if there is only 1 or no categories where the score is positive.
Berlin questionnaire | 14-18 months from baseline (after z-activator (MAD))
  The questionnaire consists of 2 categories related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories 1 and 2.
  Category 1: 5 questions. Positive score if ≥2 points Category 2: 3 questions. Positive score if ≥2 points High Risk: if there are 2 or more categories where the score is positive. Low Risk: if there is only 1 or no categories where the score is positive.

SECONDARY OUTCOMES:
Acoustic pharyngometry | Baseline
  Volumen of mouth/pharynx measured in volume cm3 Minimum cross-sectional area (MCA) measured in cm2 Distance to MCA in cm.
Acoustic pharyngometry | 4-8 months from baseline (after expansion plate)
  Volumen of mouth/pharynx measured in volume cm3 Minimum cross-sectional area (MCA) measured in cm2 Distance to MCA in cm.
Acoustic pharyngometry | 14-18 months from baseline (after z-activator (MAD))
  Volumen of mouth/pharynx measured in volume cm3 Minimum cross-sectional area (MCA) measured in cm2 Distance to MCA in cm.
Acoustic rhinometry | Baseline
  Calculated resistance (cm H2O/L/min) Volume of the nasal cavity (cm3) Minimum cross-sectional area (MCA) measured in cm2 Distance to MCA in cm.
Acoustic rhinometry | 4-8 months from baseline (after expansion plate)
  Calculated resistance (cm H2O/L/min) Volume of the nasal cavity (cm3) Minimum cross-sectional area (MCA) measured in cm2 Distance to MCA in cm.
Acoustic rhinometry | 14-18 months from baseline (after z-activator (MAD))
  Calculated resistance (cm H2O/L/min) Volume of the nasal cavity (cm3) Minimum cross-sectional area (MCA) measured in cm2 Distance to MCA in cm.
Cephalometric x-ray | Baseline
  Performed in study group before and after treatment to calculate the upper airway dimensions (cm^2).
  Margins: Superior: Hard and soft palate; Inferior: Vallecula (plane of the hyoid bone; base of the epiglottis); Anterior: Circumvallate papillae and the oropharyngeal isthmus; Posterior: Respective pharyngeal wall Results adjusted for height and weight and compared over time.
Cephalometric x-ray | 14-18 months from baseline (after z-activator (MAD))
  Performed in study group before and after treatment to calculate the upper airway dimensions (cm^2).
  Margins: Superior: Hard and soft palate; Inferior: Vallecula (plane of the hyoid bone; base of the epiglottis); Anterior: Circumvallate papillae and the oropharyngeal isthmus; Posterior: Respective pharyngeal wall Results adjusted for height and weight and compared over time.
Cone-Beam Computed Tomography | Baseline
  Performed in study group before and after treatment to calculate the upper airway dimensions (cm^3).
  Margins: Superior: Hard and soft palate; Inferior: Vallecula (plane of the hyoid bone; base of the epiglottis); Anterior: Circumvallate papillae and the oropharyngeal isthmus; Posterior: Respective pharyngeal wall; Lateral: Respective pharyngeal walls Results adjusted for height and weight and compared over time.
Cone-Beam Computed Tomography | 14-18 months from baseline (after z-activator (MAD))
  Performed in study group before and after treatment to calculate the upper airway dimensions (cm^3).
  Margins: Superior: Hard and soft palate; Inferior: Vallecula (plane of the hyoid bone; base of the epiglottis); Anterior: Circumvallate papillae and the oropharyngeal isthmus; Posterior: Respective pharyngeal wall; Lateral: Respective pharyngeal walls Results adjusted for height and weight and compared over time.

OTHER OUTCOMES:
Dental occlusion | Baseline
  3D imaging dental scanning. Width and height of the palate (mm) between upper canines and upper first molars. Results adjusted for height and weight and compared between the groups, and within the groups over time.
Dental occlusion | 4-8 months from baseline (after expansion plate)
  3D imaging dental scanning. Width and height of the palate (mm) between upper canines and upper first molars. Results adjusted for height and weight and compared between the groups, and within the groups over time.
Dental occlusion | 14-18 months from baseline (after z-activator (MAD))
  3D imaging dental scanning. Width and height of the palate (mm) between upper canines and upper first molars. Results adjusted for height and weight and compared between the groups, and within the groups over time.
Nordic Orofacial Test-Screening | Baseline
  The interview part focuses on 'sensory function', 'breathing', 'habits', 'chewing/swallowing', 'drooling' and 'dryness of the mouth'; and the examination part focuses on 'face at rest', 'nose breathing', 'facial expression', 'masticatory muscle and jaw function', 'oral motor function' and 'speech'. The NOT-S results in a score from 0 to 12; and the larger NOT-S score, the severe orofacial dysfunction and reverse.
Nordic Orofacial Test-Screening | 4-8 months from baseline (after expansion plate)
  The interview part focuses on 'sensory function', 'breathing', 'habits', 'chewing/swallowing', 'drooling' and 'dryness of the mouth'; and the examination part focuses on 'face at rest', 'nose breathing', 'facial expression', 'masticatory muscle and jaw function', 'oral motor function' and 'speech'. The NOT-S results in a score from 0 to 12; and the larger NOT-S score, the severe orofacial dysfunction and reverse.
Nordic Orofacial Test-Screening | 14-18 months from baseline (after z-activator (MAD))
  The interview part focuses on 'sensory function', 'breathing', 'habits', 'chewing/swallowing', 'drooling' and 'dryness of the mouth'; and the examination part focuses on 'face at rest', 'nose breathing', 'facial expression', 'masticatory muscle and jaw function', 'oral motor function' and 'speech'. The NOT-S results in a score from 0 to 12; and the larger NOT-S score, the severe orofacial dysfunction and reverse.
Bite force (BF) | Baseline
  BF examination done by the use of a Flöy-strand. The average of the four measurements was calculated and registered as the maximum BF in Newton (kg*m/s^2).
Bite force (BF) | 4-8 months from baseline (after expansion plate)
  BF examination done by the use of a Flöy-strand. The average of the four measurements was calculated and registered as the maximum BF in Newton (kg*m/s^2).
Bite force (BF) | 14-18 months from baseline (after z-activator (MAD))
  BF examination done by the use of a Flöy-strand. The average of the four measurements was calculated and registered as the maximum BF in Newton (kg*m/s^2).
DC/TMD | Baseline
  Symptom Questionnaire' familiar symptoms related to temporomandibular joint (TMJ), regarding five different topics: 'pain', 'headache', 'jaw joint noises', 'closed locking of the jaw' and 'open locking of the jaw', was examined. Clinical examination of jaw mobility (mm), TMJ and masticatory muscles ascertained according to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) using DC/TMD Axis I. On the basis of clinical DC/TMD examination and the questionnaire the diagnostic was made according to the DC/TMD and categorized in three groups: no TMD diagnosis, myofascial pain diagnosis and joint displacements diagnosis.
DC/TMD | 4-8 months from baseline (after expansion plate)
  Symptom Questionnaire' familiar symptoms related to temporomandibular joint (TMJ), regarding five different topics: 'pain', 'headache', 'jaw joint noises', 'closed locking of the jaw' and 'open locking of the jaw', was examined. Clinical examination of jaw mobility (mm), TMJ and masticatory muscles ascertained according to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) using DC/TMD Axis I. On the basis of clinical DC/TMD examination and the questionnaire the diagnostic was made according to the DC/TMD and categorized in three groups: no TMD diagnosis, myofascial pain diagnosis and joint displacements diagnosis.
DC/TMD | 14-18 months from baseline (after z-activator (MAD))
  Symptom Questionnaire' familiar symptoms related to temporomandibular joint (TMJ), regarding five different topics: 'pain', 'headache', 'jaw joint noises', 'closed locking of the jaw' and 'open locking of the jaw', was examined. Clinical examination of jaw mobility (mm), TMJ and masticatory muscles ascertained according to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) using DC/TMD Axis I. On the basis of clinical DC/TMD examination and the questionnaire the diagnostic was made according to the DC/TMD and categorized in three groups: no TMD diagnosis, myofascial pain diagnosis and joint displacements diagnosis.
Chew-efficiency | Baseline
  Chewing time (seconds, s) of 10 gram of a standardized Granny Smith apple slice with the rind and core removed. No normal values are previously estimated.
Chew-efficiency | 4-8 months from baseline (after expansion plate)
  Chewing time (seconds, s) of 10 gram of a standardized Granny Smith apple slice with the rind and core removed. No normal values are previously estimated.
Chew-efficiency | 14-18 months from baseline (after z-activator (MAD))
  Chewing time (seconds, s) of 10 gram of a standardized Granny Smith apple slice with the rind and core removed. No normal values are previously estimated.
Well-being | Baseline
  Strength and difficulties questionnaire examining well-being: emotional symptoms, conduct problems, inattention, peer relationship problems, prosocial behaviour. 25 questions with graduated score (true, partly true, not true).
Well-being | 4-8 months from baseline (after expansion plate)
  Strength and difficulties questionnaire examining well-being: emotional symptoms, conduct problems, inattention, peer relationship problems, prosocial behaviour. 25 questions with graduated score (true, partly true, not true).
Well-being | 14-18 months from baseline (after z-activator (MAD))
  Strength and difficulties questionnaire examining well-being: emotional symptoms, conduct problems, inattention, peer relationship problems, prosocial behaviour. 25 questions with graduated score (true, partly true, not true).
Quality of life | Baseline
  Questionnaire KIDSCREEN-10 examining quality of life 10 questions with graduating score, higher score indicate higher quality of life
Quality of life | 4-8 months from baseline (after expansion plate)
  Questionnaire KIDSCREEN-10 examining quality of life 10 questions with graduating score, higher score indicate higher quality of life
Quality of life | 14-18 months from baseline (after z-activator (MAD))
  Questionnaire KIDSCREEN-10 examining quality of life 10 questions with graduating score, higher score indicate higher quality of life
Height | Baseline
  Height without shoos in meter
Height | 4-8 months from baseline (after expansion plate)
  Height without shoos in meter
Height | 14-18 months from baseline (after z-activator (MAD))
  Height without shoos in meter
Weight | Baseline
  Weight without shoos in kilograms
Weight | 4-8 months from baseline (after expansion plate)
  Weight without shoos in kilograms
Weight | 14-18 months from baseline (after z-activator (MAD))
  Weight without shoos in kilograms
Body Mass Index | Baseline
  Body Mass Index (BMI= kg/m^2)
Body Mass Index | 4-8 months from baseline (after expansion plate)
  Body Mass Index (BMI= kg/m^2)
Body Mass Index | 14-18 months from baseline (after z-activator (MAD))
  Body Mass Index (BMI= kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Hansen, DDS, PhD student, Principal Investigator — Section of Orthodontics, Department of Odontology, University of Copenhagen
Locations (1):
- University of Copenhagen, Department of Odontology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anandarajah S, Dudhia R, Sandham A, Sonnesen L. Risk factors for small pharyngeal airway dimensions in preorthodontic children: A three-dimensional study. Angle Orthod. 2017 Jan;87(1):138-146. doi: 10.2319/012616-71.1. Epub 2016 Jun 15. PMID 27304232
- [Background] Abdalla Y, Brown L, Sonnesen L. Effects of a fixed functional appliance on upper airway volume: A 3-dimensional cone-beam computed tomography study. Am J Orthod Dentofacial Orthop. 2020 Jul;158(1):40-49. doi: 10.1016/j.ajodo.2019.07.013. Epub 2020 May 7. PMID 32389570
- [Background] Petri N, Christensen IJ, Svanholt P, Sonnesen L, Wildschiodtz G, Berg S. Mandibular advancement device therapy for obstructive sleep apnea: a prospective study on predictors of treatment success. Sleep Med. 2019 Feb;54:187-194. doi: 10.1016/j.sleep.2018.09.033. Epub 2018 Nov 12. PMID 30580193
- [Background] Andersson H, Sonnesen L. Sleepiness, occlusion, dental arch and palatal dimensions in children attention deficit hyperactivity disorder (ADHD). Eur Arch Paediatr Dent. 2018 Apr;19(2):91-97. doi: 10.1007/s40368-018-0330-3. Epub 2018 Mar 14. PMID 29542042
- [Background] Knappe SW, Sonnesen L. Mandibular positioning techniques to improve sleep quality in patients with obstructive sleep apnea: current perspectives. Nat Sci Sleep. 2018 Feb 2;10:65-72. doi: 10.2147/NSS.S135760. eCollection 2018. PMID 29440942
- [Background] Sonnesen L, Petersson A, Berg S, Svanholt P. Pharyngeal Airway Dimensions and Head Posture in Obstructive Sleep Apnea Patients with and without Morphological Deviations in the Upper Cervical Spine. J Oral Maxillofac Res. 2017 Sep 30;8(3):e4. doi: 10.5037/jomr.2017.8304. eCollection 2017 Jul-Sep. PMID 29142656
- [Background] Anandarajah S, Abdalla Y, Dudhia R, Sonnesen L. Proposal of new upper airway margins in children assessed by CBCT. Dentomaxillofac Radiol. 2015;44(7):20140438. doi: 10.1259/dmfr.20140438. Epub 2015 Mar 25. PMID 25806863
- [Background] Sonnesen L, Bakke M. Molar bite force in relation to occlusion, craniofacial dimensions, and head posture in pre-orthodontic children. Eur J Orthod. 2005 Feb;27(1):58-63. doi: 10.1093/ejo/cjh069. PMID 15743864
- [Background] Sonnesen L, Bakke M, Solow B. Malocclusion traits and symptoms and signs of temporomandibular disorders in children with severe malocclusion. Eur J Orthod. 1998 Oct;20(5):543-59. doi: 10.1093/ejo/20.5.543. PMID 9825557
- [Background] Lin SY, Su YX, Wu YC, Chang JZ, Tu YK. Management of paediatric obstructive sleep apnoea: A systematic review and network meta-analysis. Int J Paediatr Dent. 2020 Mar;30(2):156-170. doi: 10.1111/ipd.12593. Epub 2019 Nov 22. PMID 31680340
- [Background] Fagundes NCF, Flores-Mir C. Pediatric obstructive sleep apnea-Dental professionals can play a crucial role. Pediatr Pulmonol. 2022 Aug;57(8):1860-1868. doi: 10.1002/ppul.25291. Epub 2021 Mar 1. PMID 33501761
- [Background] Jennum P, Ibsen R, Kjellberg J. Morbidity prior to a diagnosis of sleep-disordered breathing: a controlled national study. J Clin Sleep Med. 2013 Feb 1;9(2):103-8. doi: 10.5664/jcsm.2398. PMID 23372461
- [Background] Knappe SW, Sonnesen L. The Reliability and Influence of Body Position on Acoustic Pharyngometry and Rhinometry Outcomes. J Oral Maxillofac Res. 2020 Dec 31;11(4):e1. doi: 10.5037/jomr.2020.11401. eCollection 2020 Oct-Dec. PMID 33598109
- [Background] Kaditis AG, Alonso Alvarez ML, Boudewyns A, Alexopoulos EI, Ersu R, Joosten K, Larramona H, Miano S, Narang I, Trang H, Tsaoussoglou M, Vandenbussche N, Villa MP, Van Waardenburg D, Weber S, Verhulst S. Obstructive sleep disordered breathing in 2- to 18-year-old children: diagnosis and management. Eur Respir J. 2016 Jan;47(1):69-94. doi: 10.1183/13993003.00385-2015. Epub 2015 Nov 5. PMID 26541535
- [Background] Ahmad M, Hollender L, Anderson Q, Kartha K, Ohrbach R, Truelove EL, John MT, Schiffman EL. Research diagnostic criteria for temporomandibular disorders (RDC/TMD): development of image analysis criteria and examiner reliability for image analysis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Jun;107(6):844-60. doi: 10.1016/j.tripleo.2009.02.023. PMID 19464658
- [Derived] Hansen C, Markstrom A, Bakke M, Sonnesen L. Sleep-Disordered Breathing and Dimensions of The Maxillary Dental Arch and Hard Palate in Children With Class II and Large Overjet-A Case-Control Study. J Oral Rehabil. 2025 Mar;52(3):367-374. doi: 10.1111/joor.13911. Epub 2024 Dec 8. PMID 39648069
- [Derived] Hansen C, Sonnesen L, Bakke M, Markstrom A. Prevalence of sleep-disordered breathing in children and adolescents with large horizontal maxillary overjet due to mandibular retrognathia: a case-control study. J Clin Sleep Med. 2024 Dec 1;20(12):1871-1878. doi: 10.5664/jcsm.11248. PMID 38958059
- [Derived] Hansen C, Sonnesen L, Markstrom A. Signal quality of home polygraphy in children and adolescents. Acta Paediatr. 2023 Dec;112(12):2583-2588. doi: 10.1111/apa.16964. Epub 2023 Sep 4. PMID 37661830
- See also: Strength and Difficulties Questionnaire — https://sdqinfo.org/a0.html
- See also: KIDSCREEN-10 — https://www.kidscreen.org/english/questionnaires/kidscreen-10-index/